CLINICAL TRIAL: NCT02823782
Title: MRI Investigations in Attention Deficit Hyperactivity Disorder (ADHD) and High Potential (HP) Children for a Better Therapeutic Approach
Acronym: HP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-805
Record Dates: First submitted 2016-06-09; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: ADHD
Keywords: Laminar HP; Complex HP
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Laminar HP (Experimental): Structural and functional MRI markers
  Interventions: Other: MRI; Other: neuropsychological assessment
- Complex HP (Experimental): Structural and functional MRI markers
  Interventions: Other: MRI; Other: neuropsychological assessment
- ADHD (Experimental): Structural and functional MRI markers
  Interventions: Other: MRI; Other: neuropsychological assessment
- Control (Other): Structural and functional MRI markers
  Interventions: Other: MRI; Other: neuropsychological assessment

INTERVENTIONS:
Other: MRI — MRI and neuropsychological assessment planned for the study for patient and volunteers
Other: neuropsychological assessment

SUMMARY:
Impulsivity and/or hyperactivity in children has become one of the main clinical symptom for consultation, among the most frequent, in general or pediatric medicine. Among the different clinical forms of instability, ADHD appears to be an especially disabling condition for the development of the child, both in psychomotor, cognitive, emotional and relational aspects. Further, a significant link between ADHD children and some children with High Potential (HP) is observed. HP children show overall ahead cognitive developments compared to children with the same age. In these children, as well as in children with ADHD, an attention vulnerability, psychomotor deficits are noted, as well as emotional and relational deficits that significantly contrasted with some of their cognitive skills. Regarding the HP, the hypothesis is that children with significantly heterogeneous results (Complex) to the Wechsler IV scales are affected by this shift, and hence, by the difficulty of a differential diagnosis with ADHD, unlike those whose intelligence quotient (IQ) results that are more homogeneous (Laminar).

The goal of this work was to study a population of 80 children aged from 8 to 12 years (20 subjects per group) to evaluate the functional and structural brain development by:

* Functional magnetic resonance imaging (fMRI) acquisitions with cognitive stimulations, involving attention, working memory and semantic processing, and emotional stimulations,
* fMRI acquisitions at rest (without activation),
* diffusion tensor magnetic resonance imaging (DTI) acquisitions,
* 3D anatomic acquisitions. Identification of developmental differences in certain cortical brain areas (eg, prefrontal vs parietal), white matter fiber bundles or functional networks preferentially used by one or other of these groups, will help to better understand this disease, and to improve the differential diagnosis in order to implement a more appropriate and personalized management of the patients via new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Right-hand 4 groups :
* Laminar HP : IQ > 130 and difference between Verbal Comprehension Index (VCI) and Perceptual Reasoning Index (PRI) < 9
* Complex HP : IQ > 130 and difference between VCI and PRI >15
* ADHD : 90 < IQ <110
* Controls : 90 < IQ <110

Exclusion Criteria:

* Subjects with any psychiatric disorders except ADHD,
* Subjects with known learning deficits (dyslexia, dysphasia…), attention deficits except for ADHD group
* Subjects with claustrophobia or magnetic devices
* Children with out both parental agreements

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Cortical gray matter (GM) volumes | Day 1
  using the software VBM (Voxel Based Morphometry)
Microstructural connectivity of white matter (WM) fiber bundles | Day 1
  measured by diffusion tensor imaging. Diffusion metrics maps are compared using the software TBSS (Track Based Spatial Statistics),
Functional MRI activity during cognitive tests | Day 1
  using the software SPM (Statistical Parametric Mapping)
Functional connectivity in resting-state fMRI | Day 1
  using the CONN toolbox (functional connectivity toolbox) of SPM (Statistical Parametric Mapping)
Subcortical gray matter (GM) volumes | Day 1
  using the software VBM (Voxel Based Morphometry)
Functional MRI activity during emotional tests | Day 1
  using the software SPM (Statistical Parametric Mapping)
Functional connectivity in resting-state fMRI | Day 1
  using the graph-theory methods

CONTACTS AND LOCATIONS:
Overall Officials: Olivier REVOL, MD, Principal Investigator — HCL
Locations (1):
- Service de psychiatrie infantile, Hôpital Pierre Wertheimer, 59 Boulevard Pinel, Bron, France